CLINICAL TRIAL: NCT02049281
Title: A Phase I Dose Escalation Study Evaluating MK-8109 (Vintafolide) in Japanese Subjects With Advanced Solid Tumor
Brief Title: A Study of Vintafolide (MK-8109) in Participants With Advanced Solid Tumor (MK-8109-011)
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Endocyte (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 8109-011; 142501 (Registry Identifier: JAPIC-CTI)
Record Dates: First submitted 2014-01-28; First posted 2014-01-30 (Estimated); Last update posted 2015-02-10 (Estimated); Status verified 2015-02

CONDITIONS: Solid Tumor
MeSH Terms: interventions — EC145

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Vintafolide (Experimental): Participants receive vintafolide intravenous (IV) bolus, starting dose 1.4 mg, on Days 1, 3, 5, 15, 17, and 19 of each 28-day cycle for up to 6 cycles.
  Interventions: Drug: Vintafolide

INTERVENTIONS:
Drug: Vintafolide — Intravenous (IV) bolus, starting dose 1.4 mg, on Days 1, 3, 5, 15, 17, and 19 of each 28-day cycle for up to 6 cycles.
  Other Names: MK-8109

SUMMARY:
This study will evaluate thrice weekly dosing with vintafolide to find the maximum tolerable dose. The primary study hypothesis is that administration of vintafolide to participants with advanced solid tumors will have acceptable safety and tolerability.

ELIGIBILITY:
Inclusion Criteria:

* Histologically-confirmed metastatic or locally advanced solid tumor that has failed to respond to standard therapy, progressed despite standard therapy, or for which standard therapy does not exist
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Adequate organ function

Exclusion Criteria:

* Chemotherapy, radiotherapy, or biological therapy (including monoclonal antibodies) within 4 weeks prior to drug administration (6 weeks for nitrosoureas or mitomycin C) or not recovered from adverse events due to agents administered more than 4 weeks earlier
* Primary central nervous system (CNS) tumor
* Active CNS metastases and/or carcinomatous meningitis
* Known hypersensitivity to the components of the study therapy or its analogs
* Recent history of abdominal surgery or peritonitis
* Bowel occlusion or sub occlusion
* Prior abdominal or pelvis radiation therapy or radiation therapy to > 10% of the bone marrow at any time in the past or prior radiation therapy within the last three years to the breast / sternum, head, or neck
* Requires anti-folate therapy
* Symptomatic ascites or pleural effusion
* Prior stem cell or bone marrow transplant

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2014-02; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Number of Participants Experiencing Dose-limiting Toxicities | Up to 28 days

SECONDARY OUTCOMES:
Maximum Plasma Concentration (Cmax) of Vintafolide | Cycle 1, Day1 predose and at 2, 5, 10, 20, 30, 45, 60, 90 and 120 minutes post-dose
Area Under the Plasma Concentration-time Curve (AUC) for Vintafolide | Cycle 1, Day1 predose and at 2, 5, 10, 20, 30, 45, 60, 90 and 120 minutes post-dose
Plasma Concentration of desacetylvinblastine hydrazide (DAVLBH) | Cycle 1, Day1 predose and at 2, 5, 10, 20, 30, 45, 60, 90 and 120 minutes post-dose

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC